CLINICAL TRIAL: NCT06108063
Title: Mitigation of Arthrofibrosis After Total Knee Arthroplasty Using Losartan
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Steadman Philippon Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2023-194
Record Dates: First submitted 2023-10-23; First posted 2023-10-30 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Knee Arthroplasty, Total
Keywords: TKA Losartan Arthrofibrosis
MeSH Terms: interventions — Losartan

STUDY DESIGN:
Intervention Model Description: prospective, randomized, double-blind, placebo controlled clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The Investigator or properly trained and delegated study team member (Physician Assistant) will write the prescription for the study medication. The subject's randomization number will be communicated directly to the Vail Health pharmacy. The Vail Health pharmacy will maintain an unblinded, de-identified randomization spreadsheet that documents group allocation for each subject. The Vail Health Pharmacy oversees and manages drug disbursement for research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Losartan (investigational) (Experimental): Losartan 12.5 mg, PO, BID, for four weeks post-TKA surgery (on Days 1 through 28, starting the day after surgery).
  Interventions: Drug: Losartan
- Placebo (control) (Placebo Comparator): Losartan Placebo 12.5 mg, PO, BID, for four weeks post-TKA surgery (on Days 1 through 28, starting the day after surgery).
  Interventions: Drug: Placebo - Losartan

INTERVENTIONS:
Drug: Losartan — 12.5 mg oral Losartan taken for 28 days total (4 week postoperative).
  Other Names: Losartan potassium
  Arms: Losartan (investigational)
Drug: Placebo - Losartan — Losartan appearance-matched Prosolv EasyTab SP placebo. 12.5 mg oral tablet taken for 28 days total (4 week postoperative).
  Other Names: Placebo Oral Tablet
  Arms: Placebo (control)

SUMMARY:
The purpose of this study is to evaluate the efficacy of Losartan use post-operatively for reducing or preventing the development of arthrofibrosis and the associated adverse impacts on clinical outcomes.

DETAILED DESCRIPTION:
This is a double-blind, randomized, placebo-controlled clinical trial proposed to evaluate the efficacy and safety of Losartan for reducing or preventing arthrofibrosis and improving patient-reported outcomes after total knee arthroplasty (TKA). Fibrosis will be evaluated over time after TKA using measures of knee range of motion and capsular thickening.

120 patients scheduled to undergo total knee arthroplasty will be recruited from the clinical practice of the Principal Clinical Investigator or his designee at The Steadman Clinic (TSC) and randomized into one of two arms (1:1).

ELIGIBILITY:
Inclusion Criteria:

1. Planned primary total knee arthroplasty of a single knee;
2. Male or female ≥ 18 years of age;
3. Capacity to personally give informed consent (consent via legally authorized representative will not be accepted) and who are willing to comply with all study-related procedures and assessments.

Exclusion Criteria:

1. Breastfeeding, pregnant, or planning to become pregnant during participation in the study;
2. Diagnosed with inflammatory or other arthritis caused by autoimmune disease affecting the study knee;
3. Previous knee arthroplasty on the study knee;
4. Previous infection affecting the study knee;
5. Planned total knee arthroplasty of contralateral knee to occur at any point during the study participation period;
6. Are hypotensive as confirmed by Principal Clinical Investigator or appropriate designee;
7. Planned lower extremity surgery (other than TKA in the study leg) for the duration of study participation;
8. Any condition other than knee osteoarthritis that significantly impairs ability to walk or perform other activities of daily living;
9. Currently taking: Losartan or other medication in the same drug class; Warfarin or related anticoagulants;
10. Opioid analgesics taken in the past 8 weeks and are not willing to discontinue these medications through the duration of the study (except as prescribed as standard of care in the immediate post-operative period);
11. Allergic to any active or inactive ingredient of Losartan;
12. Taking medication with known adverse Losartan interaction;
13. Subjects that have any medical condition, including malignancies, laboratory findings, and/or findings in the medical history or in the pre-study assessments that, in the opinion of the Investigator, constitutes a risk or contraindication for participation in the study or that could interfere with the study objectives, conduct, or evaluation, or prevent the patient from fully participating in all aspects of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-03-06 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Quantitative Ultrasound Measurement of Capsular Thickness at Lateral Retinaculum | Baseline, 6 weeks post-op, and 3 months post-op
  Thickness of knee joint capsule will be measured using quantitative ultrasound. The thickness will be measured using the distance between the two bright echoes seen on the ultrasound image that correspond to the superficial and deep edges of the capsule.
Knee Range of Motion | Baseline, 6 weeks post-op, and 3 months post-op
  Reported as degree of knee Flexion/Extension

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | From date of study drug dosing until the end of the study, an average of 3.5 months
  Occurrence of adverse events
TGF-ß multiplex immunoassay assessment of peripheral blood plasma/serum | Baseline, 10-17 days post-op, 6 weeks post-op, and 3 months post-op
  Biomarkers assessed will include quantifying secreted proteins related to inflammation, fibrosis, and senescence in the non-cellular fraction of the blood (e.g., serum and/or plasma) using commercially available immunocapture assays.
Flow cytometry immunosenescent phenotyping assessment of peripheral blood mononuclear cells | Baseline, 10-17 days post-op, 6 weeks post-op, and 3 months post-op
  Cell types measured via flow cytometry and analyzed via immunophenotype and senescent panels.
Knee Extensor Isometric Strength Assessment | Baseline, and 3 months post-op
  Assessed via handheld dynamometer and inclinometer containing a load cell that will digitally record the knee extension force.
Patient Reported Outcomes Questionnaire-Numeric Rating Scale for Knee Pain | Baseline, day of surgery, 10-17 days post-op, 6 weeks post-op, and 3 months post-op
  Scale from 1-10. Higher score represents greater knee pain.
Patient Reported Outcomes Questionnaire-Western Ontario and McMaster Universities | Baseline, and 3 months post-op
  Scale from 0-96. Higher score represents worse knee health.
Patient Reported Outcomes Questionnaire-Veteran's Rand 12-Item Health Survey | Baseline, and 3 months post-op
  Includes two subscales to calculate the total score. Higher score represents greater health. Scale standardized to a US Population mean of 50 and standard deviation of 10 points.

CONTACTS AND LOCATIONS:
Overall Officials: Johnny Huard, PhD, Principal Investigator — Steadman Philippon Research Institute; Scott Tashman, PhD, Principal Investigator — Steadman Philippon Research Institute
Locations (1):
- The Steadman Clinic, Vail, Colorado, United States

IPD SHARING:
Plan to Share IPD: No